CLINICAL TRIAL: NCT05346601
Title: A Randomized, Open-label, Single-dose, Single-center, Two-sequence, Two- Stage Phase I Trial of Chiauranib Capsule on Pharmacokinetics to Assess the Effect of High Fat Diet in Healthy Volunteers
Brief Title: Trial of Chiauranib Capsule on Pharmacokinetics to Assess the Effect of High Fat Diet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Collaborators: H & J CRO International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAR 108
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiauranib(In the fasting state) (Other): Experimental: Chiauranib Patients receive 50mg Chiauranib po only once In the fasting state and after 14 days receive 50mg Chiauranib po Only once with High Fat Diet
  Interventions: Drug: Chiauranib
- Chiauranib(In the high fat diet state) (Other): Experimental: Chiauranib Patients receive 50mg Chiauranib po only once with High Fat Diet and after 14 days receive 50mg Chiauranib po Only once In the fasting state
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — 50mg po only once

SUMMARY:
The purpose of this study is to further study the pharmacokinetic characteristics of Chiauranib Capsule in Healthy Volunteers with High Fat Diet.

DETAILED DESCRIPTION:
This study is a Randomized, Open-label, Single-dose, Single-center, two-sequence, two- stage Phase I Trial. 16 Healthy Volunteers will be enrolled and Randomized into two arms. 8 Healthy Volunteers were in each arm. Arm A：Patients receive 50mg Chiauranib po only once In the fasting state and after 14 days receive 50mg Chiauranib po Only once with High Fat Diet. Arm B: Patients receive 50mg Chiauranib po only once with High Fat Diet and after 14 days receive 50mg Chiauranib po Only once In the fasting state. During the trial, Blood samples were collected.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 18 Years to 45 Years
2. 19≤BMI≤26. Weight of male ≥50 kg and Weight of female 45 kg
3. at screening Healthy or NCS as determined by the Investigator based on physical examination, vital signs, a series of laboratory examinations（such as blood routine examination, et.al）and 12-lead electrocardiogram (ECG)
4. Healthy Volunteers have no plan to fertilize throughout treatment and for at least 6 months after study is stopped
5. Healthy Volunteers voluntarily sign informed consent
6. Able to communicate well with the Investigator, to comply with the requirements of the study

Exclusion Criteria:

1. Has known allegies to Chiauranib ,any of the excipients or Have a history of relevant atopy or drug hypersensitivity
2. Being hypertension or having risk of hypertension, or SBP≥140 mmHg, DBP ≥90 mmHg; or Being hypotension or having risk of hypotension, or SBP < 90 mmHg, DBP < 60 mmHg
3. Inability to take oral medication or having Gastrointestinal, liver and kidney diseases that affect drug absorption or metabolism within 6 months
4. Prior to random Having uncured diarrhea or having 4 or more episodes of diarrhea within 7 days prior to scheduled drug administration
5. Having any significant history of hemorrhagic disease or any history of coagulopathy
6. A history of frequent and severe infection(≥3 episodes)within the past 1 year, or a history of severe infection within 3 months prior to drug administration；
7. Ccr < 80 mL/min
8. Difficulty of venous blood collection
9. QTcF > 450 ms
10. Drug abuse within 5 years or used drug within 3 months prior to the study, or Urine drug screening is positive during screening
11. Heavy smokers(average daily smoking of more than 5 cigarettes/ day during past 3 months prior to screenig); heavy drinkers(average weekly drinking of more than 14 units of alcohol during past 6 months prior to screening, 1 unit =360 mL beer or 45 mL 40% spirits or 150 mL wine); Having Alcoholic products within 2 days prior to drug administration, or Alcohol breath test result ≥20 mg/dl
12. Ingestion of prescription drugs, OTC drug, Vitamin, dietary supplements or herbal products within 14 days prior to screening
13. Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism(CYP3A, CYP1A2 and CYP2D6)within 30 days prior to drug administration of the study medication, or Subjects who have taken any foods and drinks known to induce or inhibit hepatic drug metabolism within 7 days prior to drug administration
14. Intake of Tea, Coffee or other Caffeinated beverage(more than 8 cups, 1 cup=250 mL)within 14 days prior to drug administration, Intake of any food or beverage containing or metabolized to produce caffeine or xanthine within 48 hours prior to drug administration
15. Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication
16. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test
17. The abnormal result of C-reactive protein has clinical significance or Subjects testing positive for COVID-19
18. Vaccinated within 1 month prior to screening or plan to Vaccinate during the study
19. Females with a positive pregnancy test or Women of childbearing potential, pregnant and lactating women
20. Volunteer in any other study within 3 months prior to drug administration, or Volunteer in 3 times or more studies
21. Blood donation or lost more than 400mL blood within 3 months prior to the study, or Received blood transfusions within 1 month
22. Patients received major surgical operations within 6 months prior to screening, or plan to received surgical operation during the study
23. Extremes in food consumption practices
24. Other situations that the researchers considered unsuitable to enroll the subject

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Peak plasma concentration for Chiauranib(Cmax)
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Area under the concentration-time curve from zero to last quantificable concentration for Chiauranib (AUC0-t)
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Area under the concentration-time curve from zero extrapolated to infinity for Chiauranib（AUC0-inf）

SECONDARY OUTCOMES:
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Time to Cmax for Chiaruanib（Tmax）
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Elimination half-life（t1/2）
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Apparent clearance（CL/F）
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Apparent volume of distribution（Vd/F）
Pharmacokinetics of Chiauranib (in plasma) | up to 20 Days
  Elimination rate constant（λz）

CONTACTS AND LOCATIONS:
Overall Officials: LiYan Miao, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China